CLINICAL TRIAL: NCT01832493
Title: Sensor Optimization of CRT Response
Brief Title: Sensor Optimization of Cardiac Resynchronization Therapy Response
Acronym: SOCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOCR
Record Dates: First submitted 2013-03-20; First posted 2013-04-16 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac Resynchronization Therapy (Experimental): Patients implanted with a cardiac resynchronization therapy device
  Interventions: Device: Cardiac Resynchronization Therapy

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy — All study patients were evaluated for the optimal atrial-ventricular (AV) programmed interval using various methods.

SUMMARY:
The Sensor Optimization of Cardiac Resynchronization Therapy (CRT) Response (SOCR) Study is a multicenter, prospective, non-randomized acute feasibility study that is being conducted to determine if subcutaneous heart sounds and/or intracardiac impedance can acutely identify the optimal atrioventricular (AV) pacing intervals and optimal left ventricular (LV) electrodes in patients indicated for cardiac resynchronization therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be undergoing implant of a new or replacement/upgrade Medtronic CRT-P or CRT-D device for approved indications.
* Subject is implanted or will be implanted with an right ventricular (RV) lead that supports bipolar pacing and sensing (e.g. a bipolar pace/sense lead or a true bipolar defibrillation leads)
* Subject (or subject's legally authorized representative) must be willing to give informed consent
* Subjects must be at least 18 years of age

Exclusion Criteria:

* Subject has congenital heart disease
* Subject has a tachyarrhythmia (atrial and/or ventricular) at the time of enrollment and a cardioversion will not be attempted prior to the research procedure
* Subject has unstable coronary artery disease
* Subject cannot undergo transvenous catheterization
* Subject has a mechanical tricuspid or aortic valve prosthesis or history of significant structural tricuspid or aortic valvular disease
* Subject requires dual chamber cardiac pacing or single chamber (ventricular) pacing at rest for rate control
* Subject has a recent echocardiogram (within prior 6 months) which revealed the presence of an LV thrombus
* Subject is pregnant
* Subject is enrolled in a concurrent study that may confound the results of this study without documented pre-approval from Medtronic study manager

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SOCR Clinical Trial Leader, Study Director — Medtronic CRHF
Locations (9):
- United States (3):
  - Iowa Heart Center, Des Moines, Iowa
  - The Ohio State University, Columbus, Ohio
  - Mercy Hospital Fairfield, Fairfield, Ohio
- Canada (3):
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - Ottawa Heart Institute, Ottawa, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
- Hong Kong (2):
  - Grantham Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo H, Westphal P, Shahmohammadi M, Heckman LIB, Kuiper M, Cornelussen RN, Delhaas T, Prinzen FW. Heart sound-derived systolic time intervals for atrioventricular delay optimization in cardiac resynchronization therapy. Heart Rhythm. 2023 Apr;20(4):572-579. doi: 10.1016/j.hrthm.2022.12.031. Epub 2022 Dec 24. PMID 36574867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred from September 27, 2013 to January 28, 2016.
Pre-assignment Details: Eight patients exited the study prior to undergoing the research procedure: Four did not meet inclusion/exclusion criteria; In 2 cases, the physician deemed withdrawal medically necessary; and in 2 cases, the surgeon was unable to place the left ventricular (LV) lead.
Groups:
- Cardiac Resynchronization Therapy Patients: All study patients were evaluated for the optimal atrial-ventricular (AV) programmed interval using various methods.
Period: Overall Study
Arm/Group | Cardiac Resynchronization Therapy Patients
Started | 50
Completed | 42
Not Completed | 8
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 4
Not completed — Unable to place LV lead | 2

BASELINE CHARACTERISTICS:
Population: Patients undergoing the research procedure
Arm/Group | Cardiac Resynchronization Therapy Patients
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 30
Region of Enrollment [Number; unit: participants]
  Canada | 18
  United States | 10
  United Kingdom | 3
  Hong Kong | 11

OUTCOME MEASURES:

1. Primary Outcome: AV Interval Determination Using Impedance
Description: Current practices use the measurement LV dP/dt max to determine how the AV interval should be programmed in a CRT device. Intracardiac impedance is another method that could be used to determine the optimal AV interval. This outcome measure is the number of patients where the optimal AV interval setting as determined by intracardiac impedance agrees within one AV interval setting (30 milliseconds) of the optimal setting determined by LV dP/dt max.
Time Frame: During implant
Population: Patients with a RV tripolar intracardiac impedance measurement and a LV dP/dT max measurement for all AV intervals of interest.
Measure: Number; unit: participants
Arm/Group | Cardiac Resynchronization Therapy
Number analyzed (Participants) | 28
participants | 14

2. Primary Outcome: AV Interval Determination Using Heart Sounds
Description: Current practices use the measurement LV dP/dt max to determine how the AV interval should be programmed in a CRT device. A heart sounds measure, called S1 Amplitude Transition, is another method that could be used to determine the optimal AV interval. This outcome measure is the number of patients where the optimal AV interval setting as determined by heart sounds agrees within one AV interval setting (30 milliseconds) of the optimal setting determined by LV dP/dt max
Time Frame: During implant
Population: Patients with a RV tripolar S1 Amplitude Transition measurement and a LV dP/dT max measurement for all AV intervals of interest.
Measure: Number; unit: participants
Arm/Group | Cardiac Resynchronization Therapy
Number analyzed (Participants) | 26
participants | 11

3. Primary Outcome: Optimal Electrode Configuration Determination Using Impedance
Description: Current practices use the measurement LV dP/dt max to determine how the optimal electrode configuration for a CRT device. Intracardiac impedance is another method that could be used to determine the optimal electrode configuration. This outcome measure is the number of patients where the optimal electrode configuration setting as determined by intracardiac impedance agrees with the optimal setting determined by LV dP/dt max
Time Frame: During implant
Population: Patients with a RV tripolar intracardiac impedance measurement and a LV dP/dT max measurement for all electrode configurations of interest.
Measure: Number; unit: participants
Arm/Group | Cardiac Resynchronization Therapy
Number analyzed (Participants) | 31
participants | 8

4. Primary Outcome: Optimal Electrode Configuration Determination Using Heart Sounds
Description: Current practices use the measurement LV dP/dt max to determine how the optimal electrode configuration for a CRT device. Heart sounds, as measured by S1 Amplitude, is another method that could be used to determine the optimal electrode configuration. This outcome measure is the number of patients where the optimal electrode configuration setting as determined by heart sounds agrees with the optimal setting determined by LV dP/dt max
Time Frame: During implant
Population: Patients with a RV tripolar S1 amplitude measurement and a LV dP/dT max measurement for all electrode configurations of interest.
Measure: Number; unit: participants
Arm/Group | Cardiac Resynchronization Therapy
Number analyzed (Participants) | 28
participants | 12

ADVERSE EVENTS:
Time Frame: During implant to 26 days post-implant
Groups:
- All Enrolled Patients: Adverse events were collected and are reported for all 50 enrolled patients
Arm/Group | All Enrolled Patients
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Patients (N=50)
Device Stimulation Issue (General disorders) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 1 (1) — Allergic reaction to antibiotic
Myocardial Infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less